CLINICAL TRIAL: NCT03220048
Title: A Phase II, Repeated Dose, Double-Blinded, Randomised, Controlled Study to Examine the Prophylactic Efficacy, Safety and Tolerability of PrEP-001 in Healthy Subjects Subsequently Challenged With Influenza A/Perth/16/2009 (H3N2) Virus
Brief Title: Study Examining PrEP-001 in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hvivo (Industry)
Collaborators: Prep Biopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PrEP-CS-001
Record Dates: First submitted 2017-06-13; First posted 2017-07-18 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Influenza A H3N2
MeSH Terms: interventions — G004 compound

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A: Sentinel Group (Other): Sentinel group in which subjects received a challenge virus inoculum volume of 100uL on Day 0.
  Interventions: Other: Placebo Comparator
- Cohort B: PrEP-001 (Experimental): PrEP-001 6400μg dose administered equally over both nostrils and on 2 consecutive days, using a single dose nasal powder device, as per randomisation schedule.
  Interventions: Drug: PrEP-001
- Cohort B: Placebo (Experimental): Nasal dose of placebo Comparator equally divided over both nostrils and on 2 consecutive days, using a single dose nasal powder device, as per randomisation schedule.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: PrEP-001
  Other Names: JNJ-43260295-AAM
  Arms: Cohort B: PrEP-001
Other: Placebo Comparator
  Other Names: G-004
  Arms: Cohort A: Sentinel Group; Cohort B: Placebo

SUMMARY:
Phase 2 study, looking at the prophylactic efficacy, safety and tolerability to a repeated nasal dose of study drug after being infected with Influenza A/Perth/16/2009 (H3N2) virus.

DETAILED DESCRIPTION:
Screening took place up to 90 days before quarantine. Volunteers completed an informed consent and underwent screening assessments to determine their eligibility.

There were 2 study groups:

Cohort A: (Sentinel): determined the Challenge Virus infection rate after inoculation with Influenza Virus on Day 0. There was 12 subjects (open label, no randomisation) invited to attend Quarantine on Day -2 or -1.

Cohort B: Examined the prophylactic efficacy, safety and tolerability of PrEP-001 compared to placebo (randomised 1:1). Subjects attended on Day -4/-3, dosed with PrEP-001 or Placebo on Day -2 AND Day-1 and then challenged with virus (volume confirmed from Cohort A) on Day 0.

Volunteers remained in quarantine unit for 8 days after inoculation.

At day 28, end of study visit, volunteers seen and assessed by a study physician for well-being, on-going symptoms and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults as determined by medical history, physical examination, serology (HIV and Hepatitis B and C) and clinical laboratory tests.
* Female subjects were required to provide of a history of reliable contraceptive practice.

Exclusion criteria:

* Subjects who have a significant history of any tobacco use at any time.
* Any history or evidence of any clinically significant cardiovascular, dermatological gastrointestinal, endocrinological, haematological, hepatic, immunological, metabolic, urological, neurological, psychiatric, renal disease.
* Abnormal ECG

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Efthimiou, Study Chair — Sponsor's representative
Locations (1):
- hVIVO Services Ltd, QMB Bioenterprise building, London, United Kingdom

REFERENCES:
- [Derived] Malcolm BA, Aerts CA, Dubois KJ, Geurts FJ, Marien K, Rusch S, Van Dijck AH, Verloes R, Vingerhoets J. PrEP-001 prophylactic effect against rhinovirus and influenza virus - RESULTS of 2 randomized trials. Antiviral Res. 2018 May;153:70-77. doi: 10.1016/j.antiviral.2018.03.005. Epub 2018 Mar 19. PMID 29567461

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Started | 11 | 27 | 28
Completed | 11 | 25 | 27
Not Completed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo | Total
Number analyzed (Participants) | 11 | 27 | 28 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 27 | 28 | 66
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 11 | 23
  Male | 7 | 19 | 17 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 10 | 23 | 19 | 52
  White Irish | 0 | 0 | 1 | 1
  White Other | 0 | 2 | 1 | 3
  Mixed - White & Black Caribbean | 0 | 0 | 2 | 2
  Mixed - White & Asian | 0 | 1 | 1 | 2
  Asian or Asian British - Pakistani | 1 | 1 | 1 | 3
  Asian - Other | 0 | 0 | 1 | 1
  Black or Black British - African | 0 | 0 | 1 | 1
  Other | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 27 | 28 | 66

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: The Area Under the Curve (AUC) of Total Symptom Score From Day 1 (Post Viral Challenge) to Day 8 (Quarantine Discharge).
Description: Area Under the Curve (AUC) of total symptom scores (upper respiratory tract (URT), lower respiratory tract (LRT) and systemic viral symptoms (SVS)). Total symptom scores (from the symptom diary card) were used to calculate the AUC. The time unit used was minutes. Thus, the AUC unit is the total symptom score multiplied by the time period from first to last assessment in minutes (i.e score*mins).
  The minimum AUC value would be 0, for a subject who did not report any symptoms. The maximum AUC value is not provided as it would be theoretical only, with no real meaning in terms of severity.
  Higher scores indicate worse outcome than lower scores.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: score*mins
Groups:
- Cohort A: Sentinel Group: Sentinel group in which subjects received a challenge virus inoculum volume of 100uL on Day 0.
  Placebo Comparator
- Cohort B: PrEP-001: PrEP-001 6400μg dose administered equally over both nostrils and on 2 consecutive days, using a single dose nasal powder device, or Nasal dose of placebo Comparator equally divided over both nostrils and on 2 consecutive days, using a single dose nasal powder device, as per randomisation schedule.
  PrEP-001
- Cohort B: Placebo: Placebo Comparator
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Number analyzed (Participants) | 11 | 25 | 27
score*mins | 17956.5 (23780.83) | 4502.6 (6144.84) | 9859.6 (12215.84)

2. Secondary Outcome: Secondary Efficacy Endpoint: Symptom Scores: Peak Symptoms Score
Description: Using the scheduled protocol assessments from Day 1 to Day 8, this endpoint represented the highest total symptom score (defined as the sum of all 10 individual composite symptoms).
  The minimum value, for subjects who had no symptoms, would be 0. The maximum value would be 30.
  Higher scores indicate worse outcome than lower scores.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Cohort B: PrEP-001: PrEP-001 6400μg dose administered equally over both nostrils and on 2 consecutive days, using a single dose nasal powder device, as per randomisation schedule.
  PrEP-001
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Number analyzed (Participants) | 11 | 25 | 27
Score | 5.2 (5.88) | 1.7 (1.9) | 3.3 (3.28)

3. Secondary Outcome: Secondary Efficacy Endpoint: Incidence(s) of Illness and Infection: Viral Shedding
Description: The number of subjects with viral shedding. Viral shedding was measured by PCR, testing the nasopharyngeal swab samples.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Number analyzed (Participants) | 11 | 25 | 27
Participants | 7 | 13 | 21

4. Secondary Outcome: Secondary Efficacy Endpoint: Incidence(s) of Illness and Infection: Seroconversion
Description: The number of subjects with seroconversion. Seroconversion was measured by the ratio of Influenza A/Perth/16/2009 (H3N2) virus antibodies at follow-up versus pre-dose.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Number analyzed (Participants) | 11 | 25 | 27
Participants | 9 | 12 | 16

5. Secondary Outcome: Secondary Efficacy Endpoint: Viral Load Parameters: Area Under the Curve (AUC) of Viral Load, as Measured by Nasopharyngeal Swab RT-qPCR.
Description: Viral load data was supplied in Log10 Copies/mL. These values were used to calculate the Area Under the Curve (AUC) of Viral Load for each subject.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: mins*log10 copy number/mL
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Number analyzed (Participants) | 11 | 25 | 27
mins*log10 copy number/mL | 33021.8 (19676.07) | 23781.6 (14127.65) | 32944.4 (17059.07)

6. Secondary Outcome: Secondary Efficacy Endpoint: Total Weight of Nasal Discharge Produced Post Viral Challenge to Quarantine Discharge
Description: Total weight of nasal discharge (in grams) was calculated as the sum of mucus weights taken from Day 1 (Post viral challenge) to Day 8 (Quarantine Discharge).
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Number analyzed (Participants) | 11 | 25 | 27
grams | 26.580 (49.5158) | 3.959 (5.1349) | 13.414 (20.7986)

ADVERSE EVENTS:
Arm/Group | Cohort A: Sentinel Group | Cohort B: PrEP-001 | Cohort B: Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 10/11 | 17/27 | 21/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Sentinel Group (N=11) | Cohort B: PrEP-001 (N=27) | Cohort B: Placebo (N=28)
Alanine aminotransferase increased (Investigations) | 6 | 2 | 6
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 4
Blood cholesterol increased (Investigations) | 2 | 2 | 4
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 4
Low density lipoprotein increased (Investigations) | 2 | 0 | 3
C-reactive protein increased (Investigations) | 2 | 1 | 1
Lipase increased (Investigations) | 1 | 2 | 1
Blood fibrinogen increased (Investigations) | 0 | 1 | 2
Blood triglycerides increased (Investigations) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 2
White blood cell count increased (Investigations) | 0 | 1 | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 | 6 | 9
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 6 | 9
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Nervous system disorders (Nervous system disorders) | 4 | 1 | 1
Headache (Nervous system disorders) | 3 | 1 | 1
Infections and infestations (Infections and infestations) | 1 | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
General disorders and administration site conditions (General disorders) | 1 | 2 | 1
Pyrexia (General disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes